CLINICAL TRIAL: NCT06068712
Title: Proactive and Reactive Attention to Negative Templates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: attention; visual search; electroencephalogram (EEG)

STUDY DESIGN:
Intervention Model Description: Within-Subjects Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-Subjects Attentional Information (Experimental): All Participants receive all levels of the attentional cue (target, distractor, or neutral cue).
  Interventions: Behavioral: Attentional Cue Type

INTERVENTIONS:
Behavioral: Attentional Cue Type — Positive cue (target), negative cue (distractor), or neutral cue (baseline)

SUMMARY:
EEG Measures during Visual Search Task. In this line of research, the researchers having participants receive a positive (target) template cue, negative (distractor) template cue, or neutral (non-informative) template cue. Note: This is a re-analysis of previously collected data.

DETAILED DESCRIPTION:
When finding a search target, receiving a target cue or distractor cue can increase search efficiency compared to a neutral cue. The researchers are examining the neural basis of visual search when participants receive a positive (target) cue, negative (distractor) cue, or neutral (baseline) cue. Note: This is a re-analysis of previously collected data.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision, no history of neurological disorders

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10-11 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2015-04-02 (Actual)

PRIMARY OUTCOMES:
Button Press Reaction Time | During Testing (single day)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | During Testing (single day)
  Accuracy of responses to target item- we will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button
Proactive EEG Activity | During Testing (single day)
  Proactive (pre-search) Measures of EEG Theta Activity
Reactive EEG Activity | During Testing (single day)
  Reactive (post-search) Measures of EEG Alpha Activity

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.